CLINICAL TRIAL: NCT02441595
Title: Mindfulness Based Childbirth and Parenting Education - RCT of Effects on Parent and Child Health
Acronym: MBCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gunilla Lönnberg, M PH, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K63103043a
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Parent-Child Relations; Depression, Postpartum; Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Depression, Postpartum; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCP intervention (Experimental): The intervention involves eight 2.5 h weekly group sessions in which exercises in mindfulness are practiced and associated theory is taught to increase metacognition, emotional regulation and body awareness.
  Interventions: Behavioral: MBCP
- Control condition (Active Comparator): Participants in the control condition are being offered a standardized course in psychoprophylaxis.
  Interventions: Behavioral: Psychoprophylaxis

INTERVENTIONS:
Behavioral: MBCP — Eight weekly sessions 2,5 h and homework 30 min/day. Practicing various mindfulness meditations coupled with practical skills and theory of birthing and parenting.
  Arms: MBCP intervention
Behavioral: Psychoprophylaxis — Three sessions 3h each, and practices to do at home. Practical skills of relaxation and breathing techniques for labor as well as knowledge of birthing and parenting.
  Arms: Control condition

SUMMARY:
The purpose of this study is to explore if an intervention using Mindfulness Based Childbirth and Parenting education (MBCP) targeted to stressed pregnant women is effective in: 1) reducing prenatal stress, 2) preventing perinatal maternal mental ill-health, 3) preparing the mother for labor and 4) promoting positive infant-caregiver attachment.

DETAILED DESCRIPTION:
Sample: Pregnant women experiencing high levels of stress, and/or who previously have had periods of depression or anxiety, and/or who have had some childhood neglect, will be eligible for the study. A sample of 170 mothers and their partners recruited from antenatal clinics in Stockholm will be asked to participate. The participants in the study will be randomized to either treatment or control intervention. The study uses an experimental design with assessments at baseline and post-intervention as well as follow-ups at 3, 9 and 15 months post-partum. The intervention involves eight 2.5 h weekly group sessions in which exercises in mindfulness are practiced and associated theory is taught to increase metacognition, emotional regulation and body awareness. Participants in the control condition are being offered a standardized course in psychoprophylaxis.

Measurements - parental outcomes PSYCHOLOGICAL FUNCTIONING - 10 item Perceived Stress Scale [10]. Edinburgh Postnatal Depression Scale [11]. Positive States of Minds [12].

INTERVENTION ADHERENCE - Questions to assess intervention adherence. PHYSIOLOGICAL ASSESSMENTS - Heart Rate Variability (HRV) will be examined through ECG. The investigators hypothesize that the intervention will increase HRV in the pregnant women, thus providing an objective measure of stress. The investigators will test if women who receive the intervention during pregnancy have lower serum levels of the cytokines interleukin-6 and interleukin-10, Brain Derived Neurotrophic Factor-s, and Corticotrophin Releasing Hormone compared to the control group - physiological components that influence the fetus and are associated with immune response, hypothalamic-pituitary-adrenal axis functions, stress-related mood disorders and preterm delivery [13-16].

LABOUR - Labour records will be gathered from all participants.

Measurements - infants PHYSIOLOGICAL ASSESSMENTS - Heart Rate Variability (HRV) examined through ECG at 15 months of age. The investigators hypothesize that increased maternal HRV in the pregnancy will be associated with increased infant HRV. The investigators will also test if infants whose mothers have received the intervention have lower serum levels of the cytokines interleukin-6 and interleukin-10, Brain Derived Neurotrophic Factor-S, and Corticotrophin Releasing Hor-mone: Levels will be analyzed from PKU blood spots, routinely collected 3-4 days after birth.

INFANT SOCIAL AND EMOTIONAL FUNCTIONING - The attachment style of the infants will be assessed at age 15 months, using the standard Parent-Child Early Relational Assessment developed by Clark [17].

Data analysis: Appropriate methods will be applied to describe the sample. Hypothesis will be tested by multivariate repeated measures analysis of covariance (MANCOVA) with perceived stress as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

The study is open to pregnant women in the late second or early third trimester of pregnancy who are screened with a short questionnaire: Those who report high levels of perceived stress, and/or previous mental health issues such as depression/anxiety, and/or childhood neglect are included. Participants must also speak fluent Swedish.

Exclusion Criteria: Actively psychotic, having previous experience of mindfulness, third wave cognitive behavioral therapies, or related practices.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale 14-item | From baseline to 9 weeks (postintervention) and follow-ups when infant is 3, 9 and 12 months old
  A scale measuring perception of stressful experiences during the past month
Parent Child Early Relational Assessment | When infant is 12 months old
  Measures infant and primary caregiver attachment

SECONDARY OUTCOMES:
Change in Maternal heart rate variability | from baseline to 9 weeks (post-intervention)
  Examined through ECG
Change in Maternal serum levels of cytokines interleukin-6 and interleukin-10 | from baseline to 9 weeks (post-intervention)
Change in Maternal serum levels of Brain Derived Neurotrophic Factor-s | from baseline to 9 weeks (post-intervention)
Change in Maternal serum levels of Corticotrophin Releasing Hormone | from baseline to 9 weeks (post-intervention)
Change in Edinburgh Postnatal Depression Scale | From baseline to 9 weeks (postintervention) and follow-ups when infant is 3, 9 and 12 months old
  A 10-item scale measuring anxiety and depression
Change in Positive States of Minds | From baseline to 9 weeks (postintervention) and follow-ups when infant is 3, 9 and 12 months old
  A six-item scale measuring different positive emotional and cognitive experiences
Change in Five Facets of Mindfulness | From baseline to 9 weeks (postintervention) and follow-ups when infant is 3, 9 and 12 months old
  29-item scale measuring mindfulness
Labour records | 1 week after giving birth
  Labour records will be assessed as regards to labour complications and use of pain relief and labour induction
Infant serum levels of the cytokines interleukin-6 and interleukin-10 | At age 2-3 days
  Levels will be analyzed from dried PKU blood spots
Infant serum levels of Brain Derived Neurotrophic Factor-S | At age 2-3 days
  Levels will be analyzed from dried PKU blood spots
Infant serum levels of Corticotrophin Releasing Hormone | At age 2-3 days
  Levels will be analyzed from dried PKU blood spots
Infant Heart Rate Variability | At age 12 months
  Examined through ECG
Pregnancy Interveiw | Baseline measure
  Developed by Prof. Arietta Slade an interview concerning attachment to the expected child and the parents.

OTHER OUTCOMES:
Qualitative study of perceived experience of MBCP-intervention | When participants infant is 3-4 months old
  Individual in-depth interviews regarding the participants experiences of MBCP

CONTACTS AND LOCATIONS:
Overall Officials: Eva Nissen, Professor, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radmark L, Osika W, Wallen MB, Nissen E, Lonnberg G, Branstrom R, Henje E, Gardner R, Fransson E, Karlsson H, Niemi M. Autonomic function and inflammation in pregnant women participating in a randomized controlled study of Mindfulness Based Childbirth and Parenting. BMC Pregnancy Childbirth. 2023 Apr 10;23(1):237. doi: 10.1186/s12884-023-05528-2. PMID 37038176
- [Derived] Lonnberg G, Jonas W, Unternaehrer E, Branstrom R, Nissen E, Niemi M. Effects of a mindfulness based childbirth and parenting program on pregnant women's perceived stress and risk of perinatal depression-Results from a randomized controlled trial. J Affect Disord. 2020 Feb 1;262:133-142. doi: 10.1016/j.jad.2019.10.048. Epub 2019 Oct 30. PMID 31733457
- [Derived] Lonnberg G, Nissen E, Niemi M. What is learned from Mindfulness Based Childbirth and Parenting Education? - Participants' experiences. BMC Pregnancy Childbirth. 2018 Dec 3;18(1):466. doi: 10.1186/s12884-018-2098-1. PMID 30509218